CLINICAL TRIAL: NCT03884166
Title: MUcociliary Clearance IN Stroke
Acronym: MUCINS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other); Department of Infectiology and Pneumonology, Charite, Berlin (Unknown); University of Giessen (Other); University of Luebeck (Other); Labor Berlin - Charité Vivantes GmbH (Unknown)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: MUCINS
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Stroke, Ischemic
Keywords: Acute Ischemic Stroke; Bronchoscopy
MeSH Terms: conditions — Ischemic Stroke | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stroke
  Interventions: Diagnostic Test: bronchoscopy
- control
  Interventions: Diagnostic Test: bronchoscopy

INTERVENTIONS:
Diagnostic Test: bronchoscopy — Patients will undergo bronchoscopy to sample respiratory tissue in different heights in order to analyze mucociliary clearance

SUMMARY:
Stroke patients frequently suffer from stroke associated pneumonia. Pathophysiologically speaking, dysphagia and central nervous system (CNS)-injury induced immunosuppression largely contribute to the risk for pneumonia. In mouse models for stroke, the self-cleaning mechanisms of the lung are also affected by stroke, possibly further contributing to this risk.

The investigators designed a pilot-study to examine the structural and functional integrity of the self-cleaning mechanisms of the lung in stroke patients.

DETAILED DESCRIPTION:
Survival and functional outcome of stroke is strongly depending on the occurence of pneumonia (stroke-associated pneumonia, SAP). Early diagnose and treatment of SAP is paramount in the treatment of stroke patients. While dysphagia strongly contributes to its pathogenesis, recent years have also shown a strong risk-modulation by CNS injury induced immunosuppression, making stroke patients more susceptible to SAP. Additionally, murine models of stroke showed changes in mucociliary clearance as possible contributors to SAP. It remains unclear, whether structural integrity and mucociliary clearance of the respiratory epithel change in stroke patients, and whether these changes might contribute to the occurence of SAP.

Therefore, the investigators designed this exploratory observational pilot-study to examine the structural and functional integrity of respiratory epithel in severely affected stroke patients and correlate these findings to immune phenotyping and occurence of SAP. The investigators will conduct bronchoscopy in severely affected stroke patients to collect histological samples in order to evaluate multiple tissue predictors, as well as perform optical coherence tomography to examine ciliary kinetics in-vivo. The investigators will furthermore perform serum and plasma immune phenotyping, record occuring pneumonias and correlate these data in order to identify possible predictors of pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed consent signed by patient or legal representatives
* Acute ischemic stroke within the past 2 weeks (except the control group)
* Indication for diagnostic or therapeutic bronchoscopy

Exclusion Criteria:

* Confirmed lung malignancies or specific inflammations of the lungs
* Pneumonia (only control group)
* Autoimmune diseases of respiratory system (only control group)
* Chronic inflammatory diseases of respiratory system (only control group)
* chronic obstructive pulmonary disease (COPD) and spastic diseases of respiratory system (only control group)
* Patients being committed to psychiatric institutions or prisons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the observational cohort consists of severely affected stroke patients, which require diagnostic or therapeutic bronchoscopy, from within out academic stroke center (mostly from the interdisciplinary neurological-neurosurgical intensive care unit). The control group will consist of neurologically healthy individuals presenting for standard bronchoscopy for any reason, i.e. diagnostic exclusion of malignoma. These will be recruited from an academic pneumologic center. Our center is located in the metropolitan area of Berlin. Due to the exploratory, "pilot" characteristics of this study, there will be no targeted inclusion in terms of age or gender, but we aim for a representative sample.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mucociliary Clearance | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  - number of cilia (scanning electron microscopy)
Mucociliary Clearance | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  - activity of cilia given as frequency (in-vivo optical coherence tomography)

SECONDARY OUTCOMES:
Occurence of stroke-associated pneumonia | 7 days after stroke
  Pneumonia is defined according to the consensus recommendations (Smith et al., Stroke 2015)
Activity of autonomous nervous system | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  Concentration of Cortisol, Adrenaline and Noradrenaline in blood and heart frequency variability
Activity of immune System - Concentration of cytokines | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  Concentration of cytokines (IL-6, IL-13 and more) in blood
Activity of immune System - Concentration of inflammatory markers | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  Concentration of inflammatory markers (PCT, CRP) in blood
Activity of immune System - Expression of HLA-DR | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  Expression of Human Leukocyte Antigens (HLA)-DR on monocytes in antigens/cell
Structural changes in respiratory tissue (nasal, tracheal and bronchial) - Autophagy | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  Intensity of fluorescence of Light chain (LC) 3b protein, Aurora A and Human enhancer of filamentation (HEF)1
Structural changes in respiratory tissue (nasal, tracheal and bronchial) - Apoptosis | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  Intensity of fluorescence of TUNEL
Structural changes in respiratory tissue (nasal, tracheal and bronchial) - Increase of secretory cells | at time of bronchoscopy (within 2 weeks after acute ischemic stroke)
  Expression levels of surfactant protein, Muc5a, SPDEF, Foxa3

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- NeuroCure Clinical Research Center (NCRC), Charité, Mitte, Germany